CLINICAL TRIAL: NCT01000194
Title: Acute Fatty Acid Intervention Study
Brief Title: Acute Fatty Acid Intervention Study (AFAST)
Acronym: AFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Dutch Dairy Organization (NZO) (Other)
Responsible Party: Wageningen University, Department of human nutrition, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL19273.081.07; ABR19273
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Cardiovascular Disease; The Metabolic Syndrome
Keywords: postprandial; gene expression profiles; microarray
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- High polyunsaturated fat meal (Experimental): A high fat milkshake containing 55g of fat, mainly PUFA
  Interventions: Dietary Supplement: High fat meal
- High monounsaturated fat meal (Experimental): A high fat milkshake containing 55g of fat, mainly MUFA
  Interventions: Dietary Supplement: High fat meal
- High saturated fat meal (Experimental): A high fat milkshake containing 55g of fat, mainly SFA
  Interventions: Dietary Supplement: High fat meal

INTERVENTIONS:
Dietary Supplement: High fat meal — A high fat milkshake containing 55g of fat

SUMMARY:
The main objective of this study is to elucidate whether different dietary fatty acids (SFA, PUFA, butter fat and margarine fat) in a high fat load will have different effects on PBMC gene expression profiles. Secondary objectives are to elucidate the effects of these fat loads on individual plasma free fatty acid profiles, triglycerides and cholesterol levels.

DETAILED DESCRIPTION:
Nutrition plays a key role in the development of metabolic disorders like cardiovascular disease and the metabolic syndrome. Nutrients that can contribute to the risk of developing such diseases are fatty acids (FAs). It is known that fatty acids mediate their metabolic effects via changes in gene expression, through binding and subsequent activation of the transcription factor peroxisome proliferator-activated receptor (PPAR). In addition, it is known that unsaturated fatty acids are better ligands for PPAR than saturated fatty acids. Peripheral blood mononuclear cells (PBMC) express PPARalpha and are relatively easy to isolate from whole blood. We previously showed that the gene expression profiles of these cells can reflect free fatty acid increases during fasting. The question still remains whether dietary FA can influence gene expression in a similar way and, if so, whether different dietary FA result in different gene expression changes and subsequent activation of other pathways.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian men
* age between 18 and 30 years

Exclusion Criteria:

* Allergic to fish oil
* Allergic to margarine
* Allergic to cow milk or dairy products
* Current or recent (<4 weeks) use of fish oil supplements or more then four times fish/week; 24.35 g of EPA-DHA of fish per month (800 mg/day) as judged by the questionnaire.
* Body mass index (BMI) < 18 or > 25 kg/m2
* Urine glucose concentrations outside normal ranges (low to non-detectable)
* Fasting blood glucose outside the normal range (3 - 5.5 mmol/L)
* Tobacco smoking
* Taking medication that may influence the study results
* Received inoculations within 2 months of starting the study or planned to during the study
* Donated or intended to donate blood from 2 months before the study till two months after the study
* Diagnosed with any long-term medical condition (eg., diabetes, hemophilia, cardiovascular disease, anemia, gastrointestinal disease)
* Vegetarian

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Peripheral blood mononuclear cells (PBMC) gene expression profiles | 0, 2, 4, 6, 8 hours

SECONDARY OUTCOMES:
Plasma free fatty acid profiles | 0, 6 hours
Plasma free fatty acids | 0, 2, 4, 6, 8 hours
Plasma cholesterol | 0, 2, 4, 6, 8 hours
Plasma triglycerides | 0, 2, 4, 6, 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lydia A Afman, PhD, Study Director — Wageningen University; Michael Müller, PhD, Study Chair — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] Bouwens M, Grootte Bromhaar M, Jansen J, Muller M, Afman LA. Postprandial dietary lipid-specific effects on human peripheral blood mononuclear cell gene expression profiles. Am J Clin Nutr. 2010 Jan;91(1):208-17. doi: 10.3945/ajcn.2009.28586. Epub 2009 Nov 18. PMID 19923369